CLINICAL TRIAL: NCT00240916
Title: Ontogeny of Vaccine-Induced Measles Immunity Child Participant-6 and 9 Months
Brief Title: Ontogeny of Measles Immunity in Infants
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Hayley Altman Gans, Clinical Associate Professor, Stanford University
Other Study IDs: SU-11142008-1344; DMID Protocol #05-0039
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Measles
MeSH Terms: conditions — Measles | interventions — Measles Vaccine; Injections, Subcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Attenuvax (Measles Virus Live Vaccine, 0.5ml subcutaneous)
Biological: MMR-II (Measles-Mumps-Rubella Virus Live Vaccine, 0.5ml subcutaneous)

SUMMARY:
This is an immunogenicity study evaluating the development of the immune response of healthy infants following primary vaccination with Attenuvax at 6 or 9 months of age compared with responses in 12 month-old infants receiving MMR-II. Responses of infants receiving an early two dose measles vaccine regimen with the first dose given at 6 or 9 months followed by a second dose administered at 12 months will also be compared to infants given a single dose at 12 months of age (Table 2). The current approved regimen for measles vaccination is a first vaccination at 12-15 months and a subsequent vaccination at school entry.

A secondary endpoint of this study will be to assess the safety of measles vaccine administered as Attenuvax at 6 or 9 months of age and in an early two dose measles vaccine regimen with Attenuvax administered at 6 or 9 months followed by MMR-II at 12 months of age.

DETAILED DESCRIPTION:
This is an open-label immunogenicity and safety study of live attenuated Measles Vaccine (Attenuvax) and Measles-Mumps-Rubella (MMR-II) vaccine administered to healthy children at 6 (n=70), 9 (n=70), or 12 (n=70) months of age. Attenuvax (Measles Virus Vaccine Live, Merck & Co., Inc) and MMR-II (Measles-Mumps-Rubella Virus Vaccine Live, Merck & Co., Inc) will be delivered as 0.5 mL per dose, administered subcutaneously. Both vaccines are licensed for use in infants in the United States. MMR-II is recommended as part of the childhood immunization schedule by the AAP and ACIP, and Attenuvax is recommended for use as a single component vaccine in infants 6-11 months particularly for foreign travel and in measles outbreaks79. Infants vaccinated with Attenuvax at 6 or 9 months receive MMR-II at 12 months of age as recommended for follow-up vaccination. Immunization against measles is given as a trivalent formulation with mumps and rubella and is indicated as a primary dose at 12-15 months of age with a second dose recommended routinely at time of school entry, 4-6 years of age, but can be given at any earlier age provided that the interval between the first and second doses is at least 4 weeks .

Two hundred and ten healthy children attending the Palo Alto Medical Clinic will be recruited into one of three cohorts over a five year period. (Table 1). All children in cohort 1 and 2 (6 and 9 month old infants) will receive Attenuvax as part of their participation in this study followed by MMR-II at 12 months of age as part of their routine WCC and not as a study vaccine. Infants recruited into cohort 3, (twelve month old infants) will receive one dose of MMR-II at 12 months. All infants in the study (cohort 1, 2 or 3) are receiving MMR-II at 12 months as part of their routine childhood vaccines. The vaccination schedules is summarized in Table 1. Other immunizations as required for routine WCC will be administered simultaneously. Participation will entail 2-4 visits, 2-3 blood samples, and 1-2 immunizations and will end after the 9-18 month visit, totaling 3 to 12 months time of participation for a subject depending on cohort and if participants opt for a second follow-up blood sample.

ELIGIBILITY:
Inclusion Criteria:Subjects must meet all of the following criteria in order to be enrolled:

1. Healthy infants 6, 9, or 12 months (+ 3 weeks) of age
2. Free of obvious health problems as established by medical history and clinical examination before entering into the study
3. Parent/legal guardian willing and capable of signing written informed consent
4. Parent/legal guardian expected to be available for entire study
5. Parent/legal guardian can be reached by telephone

Exclusion Criteria:All subjects meeting any of the following exclusion criteria at baseline will be excluded from study participation:

1. Former premature infants (<36 weeks)
2. Birth weight < 2500grams
3. Significant underlying chronic illness
4. Immunodeficiency disease or immunosuppressive therapy in the participant
5. Any other condition which in the clinical judgment of the investigator might interfere with vaccine evaluation
6. Allergy to any components of the vaccine, including anaphylaxis or anyphalaxoid reaction to neomycin or eggs
7. Administration of an investigational drug
8. Blood products within 3 months of initial enrollment
9. Current febrile respiratory illness or other active febrile infection
10. Family history of congenital/hereditary immunodeficiency, unless immune competence of subject has been determined.
11. Blood dyscrasias, leukemia, lymphomas of any type or other malignant neoplasms affecting the bone marrow or lymphatic systems.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study populations include infants who are 6, 9, and 12 months of age, and healthy adults older than 18 years.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 1993-07; Primary Completion 2011-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Immune response to measles vaccine | 6 months

SECONDARY OUTCOMES:
Affect of maternal antibodies on immune response to measles vaccine. | 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Altman Gans, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation/Department of Pediatrics, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: Yes
Data is shared as requested by other investigators including raw data and summarized data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Is available